CLINICAL TRIAL: NCT06654869
Title: Laugh Against Cancer - Laughter Yoga Effect on Cancer Patients' Physiopsychological Symptoms; a Randomized Controlled Trial
Brief Title: Laughter Yoga Effect on Cancer Patients' Physiopsychological Symptoms
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Yasemin Ciraci Yasar, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ATATURKU-NRS-YCY-02
Record Dates: First submitted 2024-09-26; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Cancer; Nurse's Role; Quality of Life
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 2 (No Intervention)
- Arm 1 (Experimental): laughter yoga
  Interventions: Behavioral: lauhgter yoga

INTERVENTIONS:
Behavioral: lauhgter yoga — include laughter yoga effects on cancer patients' symptom management
  Arms: Arm 1

SUMMARY:
The universe of this study will consist of cancer patients and their relatives who are hospitalized in the medical oncology clinic of Atatürk University Research and Practice Hospital between Oct 2024 and Feb 2024. The researcher will stratify the patients in the control and intervention groups according to age and the type of treatment they receive in order to ensure homogeneity. Accordingly, the patient in each stratum will be selected from one of the labels prepared in a bag with the words "experimental" and "control" written on it and the patient will be included in the group written on the label. The patients in the control and intervention groups will not know which group they are in, but only the researcher will know who is in which group. In this way, blinding will be ensured and the study will be completed as single-blind.

DETAILED DESCRIPTION:
Sample Size Calculation:

The minimum number of people to be included in the sample was calculated by performing a power analysis. Using the "G.Power-3.1.7" program, the sample size was calculated with a test power of 0.80. As a result of the power analysis, it was determined that a total of 60 patients should be included in the control and intervention groups at α=0.05 level and 80% power. The patients to be included in the study will be randomized and assigned to the intervention (n=30) and control (n=30) groups. Volunteer acceptance for the study will begin after the acceptance of the study within the created work packages.

Data collection tools:

The data of the study will be collected in the experimental and control groups using the "Personal Information Form", "Edmonton Symptom Assesment Scale", "Herth Hope Scale" and "Life Engagement Scale".

Criteria for volunteers to be included in the study:

1. Being 18 years of age or older
2. Being diagnosed with cancer and having knowledge about the disease
3. Not having a physical illness or cognitive disability that would prevent understanding the scales used for data collection and the education provided, and not having a psychiatric illness diagnosis
4. Being literate
5. Being open to communication and collaboration

ELIGIBILITY:
Inclusion Criteria:

1. Being 18 years of age or older
2. Being diagnosed with cancer and having knowledge about the disease
3. Not having a physical illness or cognitive disability that would prevent understanding the scales used for data collection and the education provided, and not having a psychiatric illness diagnosis
4. Being literate
5. Being open to communication and collaboration

Exclusion Criteria:

1. Being under 18 years of age
2. Not having information about the disease
3. Having a physical illness or cognitive disability that prevents understanding the scales used for data collection and the education given, and being diagnosed with a psychiatric disease
4. Being illiterate
5. Not being open to communication and cooperation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Edmonton Symptom Assesment Scale (ESAS) | 6 weeks
  Bruera et al. (1991) to evaluate nine symptoms commonly seen in cancer patients. These symptoms are pain, fatigue, nausea, sadness, anxiety, insomnia, loss of appetite, feeling good, shortness of breath and other problems. In the other problems section of the scale, 2 additional symptoms seen in patients by researchers (feeling of thirst and discomfort due to catheters and catheters) were added in accordance with literature information. The severity of each symptom is evaluated with numerical numbers from 0 to 10. A score of 0 indicates that there is no symptom, a score of 10 indicates that the symptom is felt very severely, and the severity of the symptom increases from 0 to 10.
Life Engagement Scale | 6 weeks
  The Life Engagement scale, developed by Scheier et al. (2006) to assess individuals' life goals and whose Turkish validity and reliability were determined by Akın et al., is a measurement tool consisting of 6 items and a single dimension (life engagement). The scale has a 5-point scale ("1" I completely disagree, "5" I completely agree). Items 1, 3 and 5 are reverse coded in the scale. Increasing scores indicate a high level of life engagement.
Herth Hope Scale | 6 weeks
  The Herth Hope Scale was developed by Kaye Herth. The scale consists of 30 items. Each item has four options: "Never " "Rarely appropriate," "Sometimes" and "Always " . The corresponding scores are 0, 1, 2, and 3, respectively. The respondent is asked to mark a single option for each item. The scale consists of 3 sub-dimensions. These are "Future," "Positive Readiness and Expectation," and "Relationships Between Oneself and Those Around Oneself." The "Future" sub-dimension measures the cognitive-temporal dimension of hope, the "Positive Readiness and Expectation" sub-dimension measures the emotional-behavioral dimension of hope, and the "Relationships Between Oneself and Those Around Oneself" sub-dimension measures the dimension of hope related to relationships and the conditions in which it exists. The total hope score varies between 0-90, and the total score of each subscale varies between 0-30. High scores, It shows that hope is high.

IPD SHARING:
Plan to Share IPD: Undecided